CLINICAL TRIAL: NCT01160406
Title: Improving Screening for Silent Atrial Fibrillation, After Ischemic Stroke
Brief Title: Screening for Atrial Fibrillation, After Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Mårten Rosenqvist M.D. Ph.D., Karolinska Institutet
Other Study IDs: KI-DSAB-2010
Record Dates: First submitted 2010-07-09; First posted 2010-07-12 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: silent paroxysmal atrial fibrillation; stroke; tele ECG
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ischemic stroke, no atrial fibrillation: Patients who have suffered ischemic stroke or transient ischemic attack without known atrial fibrillation

SUMMARY:
The aim of the study is to assess the incidence of patients suffering from ischemic stroke or transient ischemic attacks who have underlying asymptomatic paroxysmal atrial fibrillation.

Patients who have suffered an ischemic stroke or transient ischemic attack, without a history of atrial fibrillation, are planned to be included. Starting within 14 days of the ischemic stroke, participating patients are asked to perform 10 second ECG recordings using a handheld ECG device twice daily (mornings and evenings) during 30 days. These recordings are transmitted via telephone to a secure encrypted Internet site. Within these 30 days the participants also perform an ambulatory 24 hour Holter recording. Handheld ECG recordings are evaluated continuously. In case of atrial fibrillation the patient is informed and offered treatment with anti coagulant medication (Warfarin). The investigation is a comparison between 24 hour continuous ECG recordings and short intermittent ECG recordings twice daily over a longer time period to determine which method is the best to detect atrial fibrillation in this patient group.

Hypothesis: Short Intermittent ECG recordings over a longer time period is more efficient, compared with continuous 24 hour ECG recordings, in detecting silent paroxysmal AF in patients with an ischemic stroke and without a history of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* No previously diagnosed atrial fibrillation.
* Acute ischemic stroke or transient ischemic attack verified by computed tomography or clinical diagnosis using the National Institute of Health Stroke Score within 14 days of enrollment.
* Ability to understand study instructions both verbal and written.
* Ability to perform and transmit ECG recordings according to study design.

Exclusion Criteria:

* Previously diagnosed atrial fibrillation.
* Hemorrhagic stroke
* Low compliance
* Pacemaker carrier

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from hospital strokewards.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2007-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mårten Rosenqvist, M.D.Ph.D., Study Director — Karolinska Institutet
Locations (3):
- Sweden (3):
  - Halmstad hospital, Halmstad, Halland County
  - South hospital, Stockholm, Stockholm County
  - Danderyds hospital AB, Stockholm, Stockholm County